CLINICAL TRIAL: NCT05837780
Title: Three Dimensional Evaluation of Maxillary Arch Changes After Using Two Different Construction Techniques of Nasoalveolar Molding Devices in Unilateral Cleft Lip and Palate Patients (Randomized Controlled Trial)
Brief Title: Effect of Using Two Different Construction Techniques of Nasoalveolar Molding Devices in Unilateral Cleft Lip and Palate Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Amany Alaa Abd el Aziz, assistant Lecturer of prosthodontics, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Clp04042024
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Unilateral Cleft Lip and Palate
MeSH Terms: interventions — Palatal Obturators

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventionally constructed nasoalveolar molding devices (control group) (Experimental): control group: patients receiving conventionally constructed nasoalveolar molding devices
  Interventions: Other: Nasoalveolar molding device
- Digitally constructed nasoalveolar molding devices (test group) (Experimental): test group: patients receiving digitally constructed nasoalveolar molding devices
  Interventions: Other: Nasoalveolar molding device

INTERVENTIONS:
Other: Nasoalveolar molding device — comparison between using conventionally and digitally constructed nasoalveolar molding devices

SUMMARY:
This study includes Three Dimensional Evaluation of Maxillary Arch Changes After Using Two Different Construction Techniques of Nasoalveolar Molding Devices in Unilateral Cleft Lip and Palate Patients (Randomized Controlled Trial) Null hypothesis: there is no difference between using conventionally constructed nasoalveolar molding device and using digitally constructed nasoalveolar molding device

ELIGIBILITY:
Inclusion Criteria:

Good general health without any systematic disease, disability or other syndromes Non syndromatic unilateral cleft lip and palate Both genders Age less than one month Parents willing to participate in the study and sign informed consent

Exclusion Criteria:

* Patients exhibiting systemic disease, disability or other syndrome, parents denying participating in the study or not given their informed consent

Ages: 7 Days to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Alveolar cleft width | 3 months
  measurement of width between two alveolar segments

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry ,Minya university, Minya, Egypt